

## Active Surveillance for Low-Risk Prostate Cancer -Evaluation of the Efficacy of Minimally Invasive Active Surveillance

## STHLM3 AS

## **Informed consent**

**Principal Investigator** Anna Lantz, MD PhD

## **Co-investigators in alphabetical order:**

Jan Adolfsson, MD PhD Martin Eklund, PhD Professor Henrik Grönberg, MD PhD Fredrik Jäderling, MD PhD Tobias Nordström, MD PhD Henrik Olsson, MSc

May 2019









| Informed Consent |
|------------------|

I agree to participate in STHLM 3-AS

I have read the written information about STHLM3 AS Study, or it has been read to me. I have had the opportunity to ask questions about it and any questions that I have asked have been answered to my satisfaction. I consent voluntarily to participate as a participant in this research.

I allow STHLM3 AS to process my personal information according to the information I have read, save answers to questionnaires and store my blood samples in a biobank. I allow STHLM3 AS to have access to my medical records and use information from these for health-related research that has approval from an ethics testing committee - also for research outside Sweden and the EU / EEA. I allow STHLM3 AS to obtain information about me from public records and quality registers, according to the specific information I received in the written material.

| Signature | |
|----------------------------------|------|
| Personal number and Printed name | Date |

Leave your written consent at the time of magnetic camera examination, see the first page of this letter.

If you have any questions, please do not hesitate to contact STHLM3 by phone +46 8 524 86 797 or by email sthlm3@ki.se.